CLINICAL TRIAL: NCT06924840
Title: A Clinical Evaluation of the Safety, In-Use Tolerability, and Efficacy of the Utixira Lotion and Utixira Tablet Combination Regimen in Healthy Adults With Dry, Sensitive Skin Prone to Mild to Moderate Pruritus and Urticaria
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Utixira Lotion and Utixira Tablet in Healthy Adult Human Subjects With Dry or Sensitive Skin Prone to Mild to Moderate Pruritus and Urticaria
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SAVA Healthcare Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB250006-SG
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Dry Skin; Urticaria; Pruritus; Sensitive
MeSH Terms: conditions — Urticaria; Pruritus; Hypersensitivity | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Utixira Lotion and Tablet Mode of Usage: To be applied over the affected areas twice a day as a thin film and rubbed in gently and completely. take 1 tablet twice a day for better results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Utixira Lotion tablet as regimen (Experimental): Mode of Usage: To be applied over the affected areas twice a day as a thin film and rubbed in gently and completely. take 1 tablet twice a day for better results.
  Marketed By: SAVA Healthcare Ltd Frequency: Twice a Day
  Interventions: Other: Utixira Lotion tablet as regimen

INTERVENTIONS:
Other: Utixira Lotion tablet as regimen — Mode of Usage: To be applied over the affected areas twice a day as a thin film and rubbed in gently and completely. Take 1 capsule twice a day for better results.
  Marketed By: SAVA Healthcare Ltd Frequency: Twice a Day

SUMMARY:
This exploratory, prospective, open-label, single-centre, safety, efficacy and in-use tolerability study of the Utixira Lotion + Utixira Lotion as regimen in healthy adult human subjects with dry or sensitive skin and prone to mild to moderate pruritus or urticaria

DETAILED DESCRIPTION:
A total of up to 32 healthy male and non-pregnant | non-lactating female (21 subjects with dry or sensitive skin and 11 subjects of pruritus/urticaria patients) and an age of 18-55 years will be enrolled to complete the 30 subjects the study (20 subjects with dry or sensitive skin and 10 subjects of pruritus/urticaria patients).

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called telephonically by the recruiting department prior to the enrolment visit. Subjects will be told during screening (prior to enrolment) not to wear any facial make-up on the study visit day. The adult female subjects will be instructed to visit the facility as per the below visits.

* Visit 01 (Day 01): Screening, Enrollment, Baseline Evaluation, On Site Product Usage, Post Usage Evaluation
* Visit 02 (Day 15 +2 Days): Evaluations, Product usage period
* Visit 03 (Day 30 +2 Days): Evaluations, End of the Study

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 55 years (both inclusive) at the time of consent.
* Sex: Healthy male and non-pregnant/non-lactating females.
* Females of childbearing potential must have a self-reported negative pregnancy test.
* Subject are generally in good health.
* Subject with dry or sensitive skin at a time of screening. (Dermatological Assessment)
* Subjects having pruritus or urticaria at a time of screening.
* Subjects application site must be free of cuts, tattoos, scratches, abrasions, scars, uneven skin tone, sunburn, excessive tan, excessive hair or open wounds.
* Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
* If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
* Subjects are willing to give written informed consent and are willing to come for regular follow up.
* Subjects who commit not to use medicated skincare product other than the test product for the entire duration of the study.
* Subject who have not participated in a similar investigation in the past three months.
* Willing to use test product throughout the study period.

Exclusion Criteria:

* History of any dermatological condition of the skin diseases.
* Subject with present condition of allergic response to any cosmetic product.
* Subject having allergic response to the ink.
* Presence of any broken, chapped, cut, irritated, or scraped skin at the application site.
* Subjects under chronic medication (e.g. aspirin-based products, anti-inflammatories, anti-histamines, corticotherapy etc.) that might influence the outcome of the study.
* Subject having acne of severe incidence (presence of nodules, cysts or numerous pustules) which requires pharmaceutical or cosmeceuticals, herbal treatment.

Subjects who have applied topical treatment for at least 4 weeks and any systemic treatment for at least 3 months, before they participated in the study.

* History of alcohol or drug addiction.
* Subjects using other marketed products during the study period.
* Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
* Pregnant or breastfeeding or planning to become pregnant during the study period.
* History of chronic illness which may influence the cutaneous state.
* Subjects participating in other similar cosmetics, devices or therapeutic trials or skincare products within the last four weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
1. To evaluate the effectiveness of the test product in terms of change in Urticaria | after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  UAS7 scoring scale where 0= urticaria free and 28-42 = severe urticaria
2. To evaluate the effectiveness of test product in terms of change in skin Pruritus (itching) | From baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  VAS scale where 0 = No pruritus (itching) and 10= very severe pruritus (itching)
3. To assess the effectiveness of test product in terms of change in skin hydration | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  Instrumental Evaluation: Corneometer CM 825
4. To assess the effectiveness of the test product in terms of change in DASI (Dry area and severity index) score | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  Scoring Scale: 0: absent, 4: extreme
5. To assess the effectiveness of the test product in terms of change in overall dry skin score | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  Scoring Scale: 0: absent, 4: Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks
6. To evaluate the effectiveness of the test product in terms of change in skin barrier function | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  Instrumental Evaluation: TEWAMeter TM Hex
7. To evaluate the effectiveness of the test product in terms of change in skin roughness | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  Instrumental Evaluation: VISIOSCAN VC 20 Plus
8. To evaluate the effectiveness of the test product in terms of change in skin scaliness | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  Instrumental Evaluation: VISIOSCAN VC 20 Plus
9. To evaluate the effectiveness of the test product in terms of change in skin smoothness | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  Instrumental Evaluation: VISIOSCAN VC 20 Plus
10. To evaluate the effectiveness of the test product in terms of change in skin wrinkles | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  Instrumental Evaluation: VISIOSCAN VC 20 Plus

SECONDARY OUTCOMES:
To assess the effectiveness of the test product in terms of change in redness score | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  VAS scale where 0 = No redness and 10= very severe redness
To assess the effectiveness of the test product in terms of change in visual assessment of skin dryness | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  0= Absent 4= extreme
To assess the effectiveness of the test product in terms of change in visual assessment of skin roughness | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  0= Absent 4= extreme
To assess the effectiveness of the test product in terms of change in visual assessment of skin redness | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  0= Absent 4= extreme
To assess the effectiveness of the test product in terms of change in visual assessment of ski itchiness | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  0= none 4= severe
To assess the effectiveness of the test product in terms of change in visual assessment of skin scaliness | from baseline before usage of the test product on Day 01 and after usage of the test product at T2 hours on Day 01, Day 15 (+2 Days), and Day 30 (+2 Days)
  0= Absent 4= extreme

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Principal Investigator — NovoBliss Research Private Limited

IPD SHARING:
Plan to Share IPD: No